CLINICAL TRIAL: NCT05014126
Title: Online "Pain, Stress & Emotions" Class in Chronic Pain: Single-arm Efficacy Test
Brief Title: Online "Pain, Stress & Emotions" Class in Chronic Pain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Maisa Ziadni, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: StanfordClass
Record Dates: First submitted 2021-08-12; First posted 2021-08-20 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Uncontrolled, prospective, single arm, pre-post intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain, Stress, & Emotions Class (Experimental): No active or placebo comparator will be used. This is a single-arm study design.
  Interventions: Behavioral: Pain, Stress and Emotions

INTERVENTIONS:
Behavioral: Pain, Stress and Emotions — 2-hour, zoom-delivered, group intervention focused on teaching patients how pain is processed in their brain and learning about the role of psychosocial factors in their pain conditions.

SUMMARY:
Members with chronic pain will be invited to participate in a 2-hour zoom-delivered pain psychology class entitled "Pain, Stress, & Emotions". Surveys are completed at baseline (prior to the online class), a satisfaction survey is completed after the class, and post-treatment surveys completed 2, 4, 8, and 12 1weeks after class attendance.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain condition (pain > 3 months)
* Access to the internet
* English fluency

Exclusion Criteria:

* Ongoing legal action or disability claim
* Cognitive impairment, non-English speaking, or psychological factors that would preclude comprehension of material and/or full participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Pain Intensity NRS | Change from baseline to 1-Month follow-up (with secondary 2-month follow-up)
  Self-reported pain intensity rating

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System: Pain Interference short form 6a | Change from baseline to 1-Month follow-up (with secondary 2-month follow-up)
  self-reported pain interference levels
Patient-Reported Outcomes Measurement Information System: Depression 6a | Change from baseline to 1-Month follow-up (with secondary 2-month follow-up)
  self-reported depression
Patient-Reported Outcomes Measurement Information System: Anxiety 6a | Change from baseline to 1-Month follow-up (with secondary 2-month follow-up)
  self-reported anxiety
Patient-Reported Outcomes Measurement Information System: Physical Function 8b | Change from baseline to 1-Month follow-up (with secondary 2-month follow-up)
  self-reported physical functioning
Patient-Reported Outcomes Measurement Information System: Sleep Disturbance 6a | Change from baseline to 1-Month follow-up (with secondary 2-month follow-up)
  self-reported sleep disturbance
Patient-Reported Outcomes Measurement Information System: social isolation 6a | Change from baseline to 1-Month follow-up (with secondary 2-month follow-up)
  self-reported social isolation
Patient-Reported Outcomes Measurement Information System: fatigue 6a | Change from baseline to 1-Month follow-up (with secondary 2-month follow-up)
  self-reported fatigue
Patient-Reported Outcomes Measurement Information System: anger 5a | Change from baseline to 1-Month follow-up (with secondary 2-month follow-up)
  self-reported anger
Ambivalence over Emotional Expression (AEQ) | Change from baseline to 1-Month follow-up (with secondary 2-month follow-up)
  self-reported ambivalence levels about emotional expression
Emotion-Approach Coping | Change from baseline to 1-Month follow-up (with secondary 2-month follow-up)
  8-item emotion approach coping scale
Pain Bothersomeness | Change from baseline to 1-Month follow-up (with secondary 2-month follow-up)
  single-item assessing self-reported levels of pain bothersomeness

OTHER OUTCOMES:
Pain Attributions Questionnaires | Change from baseline to 1-Month follow-up (with secondary 2-month follow-up)
  Two self-report questionnaires were developed to assess psychological and brain influences on pain. The 4-item psychological attribution scale assesses patients' beliefs that their thoughts and feelings and psychological therapy impacts pain, and the 3-item brain attribution scale assesses patient's beliefs that their pain is brain-based. Mean scores will be computed for both scales separately (0-4; higher scores indicating greater belief that pain is a brain-related [brain attribution] construct and that pain is affected by thoughts, feelings, and psychological interventions [psychological attribution])
Pain Catastrophizing Scores; measured with Pain Catastrophizing Scale | Change from baseline to 1-Month follow-up (with secondary 2-month follow-up)
  Pain Catastrophizing Scale (Sullivan et al., 1995): A summed score of the 13 catastrophizing items will be computed (0-52, higher scores indicate greater catastrophizing)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmes HJ, Thakur ER, Carty JN, Ziadni MS, Doherty HK, Lockhart NA, Schubiner H, Lumley MA. Ambivalence over emotional expression and perceived social constraints as moderators of relaxation training and emotional awareness and expression training for irritable bowel syndrome. Gen Hosp Psychiatry. 2018 Jul-Aug;53:38-43. doi: 10.1016/j.genhosppsych.2018.05.002. Epub 2018 May 3. PMID 29751205
- [Background] Carty JN, Ziadni MS, Holmes HJ, Tomakowsky J, Peters K, Schubiner H, Lumley MA. The Effects of a Life Stress Emotional Awareness and Expression Interview for Women with Chronic Urogenital Pain: A Randomized Controlled Trial. Pain Med. 2019 Jul 1;20(7):1321-1329. doi: 10.1093/pm/pny182. PMID 30252113
- [Background] Ziadni MS, Carty JN, Doherty HK, Porcerelli JH, Rapport LJ, Schubiner H, Lumley MA. A life-stress, emotional awareness, and expression interview for primary care patients with medically unexplained symptoms: A randomized controlled trial. Health Psychol. 2018 Mar;37(3):282-290. doi: 10.1037/hea0000566. Epub 2017 Nov 20. PMID 29154608
- [Background] Thakur ER, Holmes HJ, Lockhart NA, Carty JN, Ziadni MS, Doherty HK, Lackner JM, Schubiner H, Lumley MA. Emotional awareness and expression training improves irritable bowel syndrome: A randomized controlled trial. Neurogastroenterol Motil. 2017 Dec;29(12):10.1111/nmo.13143. doi: 10.1111/nmo.13143. Epub 2017 Jun 22. PMID 28643436
- [Derived] Ziadni MS, Sturgeon JA, Lumley MA. "Pain, Stress, and Emotions": Uncontrolled trial of a single-session, telehealth, emotional awareness and expression therapy class for patients with chronic pain. Front Pain Res (Lausanne). 2022 Nov 18;3:1028561. doi: 10.3389/fpain.2022.1028561. eCollection 2022. PMID 36466215